CLINICAL TRIAL: NCT07228234
Title: Evaluating Mammography Communication Approaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 25-0635; R37CA254926 (NIH)
Record Dates: First submitted 2025-11-11; First posted 2025-11-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: The Focus of This Study is to Identify How Different Approaches to Mammography Communication Affect Skepticism Toward Mammography Evidence
Keywords: Communication; Mammography
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This is a 2 x 2 +1 randomized factorial design. Participants will be randomly assigned to 1 of 5 experimental conditions, which vary (1) whether screening outcomes are referred to as "benefits and harms" vs. "outcomes that can happen with screening", and (2) the presence or absence of information about improvements in breast cancer treatment and survivability. In a 5th arm, a control condition, participants receive basic information about what mammography is (which is also information received in all other conditions).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control condition (Experimental): Participants receive basic information about what mammography screening is
  Interventions: Other: No intervention
- Harm/benefit language, survivability information (Experimental): Outcomes of screening are referred to as "harms" and "benefits"; information about breast cancer survivability is included
  Interventions: Other: Harm/benefit language vs. outcomes that can happen; Other: Breast cancer survivability information
- Harm/benefit language, no survivability information (Experimental): Outcomes of screening are referred to as "harms" and "benefits"; information about breast cancer survivability is not included
  Interventions: Other: Harm/benefit language vs. outcomes that can happen
- Outcomes that can happen language, survivability information (Experimental): Outcomes of screening are referred to as "outcomes that can happen"; information about breast cancer survivability is included
  Interventions: Other: Harm/benefit language vs. outcomes that can happen; Other: Breast cancer survivability information
- Outcomes that can happen language, no survivability information (Experimental): Outcomes of screening are referred to as "outcomes that can happen"; information about breast cancer survivability is not included
  Interventions: Other: Harm/benefit language vs. outcomes that can happen

INTERVENTIONS:
Other: Harm/benefit language vs. outcomes that can happen — Information about mortality benefit, false positives and overdiagnosis are referred to throughout the communication as either "harms" and "benefits" or "outcomes that can happen".
  Arms: Harm/benefit language, no survivability information; Harm/benefit language, survivability information; Outcomes that can happen language, no survivability information; Outcomes that can happen language, survivability information
Other: Breast cancer survivability information — Information about improvements over time in the survivability of breast cancer is provided vs. not
  Arms: Harm/benefit language, survivability information; Outcomes that can happen language, survivability information
Other: No intervention — This is the control condition in which only basic information about mammography screening.
  Arms: Control condition

SUMMARY:
This is a randomized online experiment testing different methods for communicating about the benefits and harms of breast cancer screening. Participants will be randomly assigned to experimental conditions which vary whether screening outcomes are referred to as "benefits and harms" vs. "outcomes that can happen with screening", and vary the presence or absence of information about improvements in breast cancer survivability. In a control condition, participants receive basic information about what mammography is (which is also information received in all other conditions). Primary outcomes include skepticism toward the information presented, and screening intentions.

DETAILED DESCRIPTION:
This is a randomized online experiment testing different methods for communicating about the benefits and harms of breast cancer screening. Participants will be randomly assigned to 1 of 5 experimental conditions, in a 2 x 2 + 1 factorial design, which vary (1) whether screening outcomes are referred to as "benefits and harms" vs. "outcomes that can happen with screening", and (2) the presence or absence of information about improvements in breast cancer treatment and survivability. In a 5th arm, a control condition, participants receive basic information about what mammography is (which is also information received in all other conditions). Primary outcomes include skepticism toward the information presented, and screening intentions.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 39-49

Exclusion Criteria:

* No history of breast cancer, no known BRCA1/2 gene mutation

Ages: 39 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1900 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Skepticism toward the screening message | Participant experience entails a one-time survey. This outcome is measured in that survey, immediately after participants read information about mammography screening.
  Skepticism toward the screening message is assessed using the RED scale, consisting of 11 questions each measured on a 7-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Although these data are anonymized, data will be checked for any potentially identifying information. Any such information will be removed from the data prior to data sharing. The full data (sans potential identifiers) will be made publicly available on the Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: This information will be made publicly available on the Open Science Framework prior to publishing the a manuscript from these data.
Access Criteria: Anyone will be able to access the IPD via the Open Science Framework.
URL: https://osf.io/6m4y8/overview